CLINICAL TRIAL: NCT06451835
Title: Evaluation of Response to a Course of Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Major Depressive Disorder Using Vocal Biomarkers
Brief Title: Evaluation of Response to a Course of Repetitive Transcranial Magnetic Stimulation Using Vocal Biomarkers
Acronym: SPEECHTMS
Status: Suspended | Type: Observational
Why Stopped: We are faced with a decrease in rTMS activity at the study sites, as well as problems with the active file meeting the protocol inclusion criteria, resulting in a low recruitment rate and an extended study timetable, forcing us to suspend this study.
Sponsor: GCS CIPS (Other)
Collaborators: Callyope (Industry)
Responsible Party: Sponsor
Other Study IDs: SPEECHTMS
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with MDD: Patients who are prescribed a course of 30 rTMS sessions to treat an episode of MDD at one of the nine participating centres
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — rTMS will be applied 5 days out of 7 for 6 weeks, for a total of 30 sessions. The area stimulated will be the left dorsolateral prefrontal cortex, at a frequency of 10 Hz, at 110% of motor threshold for approximately 20 minutes (i.e. 3,000 stimulations per session).

SUMMARY:
Voice recordings taken prior to the start of repetitive transcranial magnetic stimulation (rTMS) therapy will be used to develop a predictive model of treatment response using machine learning for patients with major depressive disorders (MDD).

DETAILED DESCRIPTION:
The objective of this study is to investigate whether voice biomarkers taken prior to the start of rTMS can predict the response to a 30-session course of rTMS in patients with MDD with good sensitivity and specificity. Patients who are prescribed rTMS to treat an episode of MDD at one of the nine participating centres will be invited to participate in the study. The protocol includes one inclusion visit and seven evaluation visits before, during, and after the course of rTMS. The rTMS course will last for six weeks, comprising of 30 sessions with five sessions per week. Prior to the commencement of the rTMS course, patients will need to complete several questionnaires. Before the first session, voice tests will be recorded using the Callyope application. Patients will answer questionnaires and assess voice tests weekly and after the final rTMS session to track the progression of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Having a prescription for a course of rTMS to treat an episod of MDD
* Unipolar MDD confirmed according to DSM-5 criteria
* Moderate to severe MDD (MADRS score > 19)
* No use of psychotropic medication or use stabilised (no change in dose < 4 weeks before study entry)
* Able to understand, speak, read and write French
* Express informed consent, after a period of reflection
* Affiliated with a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* History of epilepsy or convulsive seizures
* Previous brain surgery
* History of recent cranial trauma (< 6 months)
* Presence of severe suicidal ideation
* Psychotic disorders
* Metal objects in the head, eyes or brain
* Implanted ferromagnetic equipment (pace maker, cochlear implant, etc.)
* Clinical evidence of serious or uncontrolled alcohol or substance use disorders in the three months prior to the study
* Active withdrawal from alcohol or other substances
* One or more recent rTMS sessions (< 4 weeks)
* Other non-drug therapy recently initiated (< 4 weeks) to treat EDC (psychotherapy, phototherapy, vagus nerve stimulation, etc.)
* Pathology altering phonation based on the perception of the investigator
* Subjects in a period of relative exclusion from another protocol
* Adults protected by law or patients under guardianship or curatorship
* Subjects deprived of their liberty by judicial or administrative decision
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients recruited will be patients admitted as outpatients to treat MDD through a rTMS treatment in one of the 9 investigation centers.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of the model predicting response to rTMS treatment | 6 weeks : before the first session of rTMS (vocal samples) and before and after the rTMS treatment (MADRS score)
  Area under the curve of the model predicting response to rTMS treatment, objectified by a 50% reduction in MADRS depression score, trained from vocal biomarkers recorded before rTMS treatment.

SECONDARY OUTCOMES:
Area under the curve of the rTMS remission prediction model | 6 weeks : before the first session of rTMS (vocal samples) and before and after the rTMS treatment (MADRS score)
  Area under the curve of the rTMS remission prediction model, objectified by a post-course MADRS score lower than 10, trained from vocal biomarkers recorded before the rTMS course.
Area under the curve of the prediction model of the self-assessed response to the rTMS course | 6 weeks : before the first session of rTMS (vocal samples) and each week during the rTMS treatment (PHQ-9 score)
  Area under the curve of the prediction model of the self-assessed response to the rTMS course, objectified by a 50% reduction in PHQ-9 depression score, trained from the vocal biomarkers recorded before the rTMS course.
Area under the curve of the prediction model of the response to the rTMS course, trained with the addition of weekly recorded voice samples. | 6 weeks : weekly
  Area under the curve of the prediction model of the response to the rTMS course, trained with the addition in the initial model of vocal biomarkers recorded each week of the rTMS course.
Area under the curve of the model predicting the response to rTMS treatment, trained with the addition of clinical indicators | 6 weeks : before the first session of rTMS (vocal samples) and before and after or weekly (clinical indicators)
  Area under the curve of the model predicting the response to rTMS treatment, trained with the addition in the initial model of clinical indicators other than depression.
Comparison between the scores predicted by the model and the actual scores obtained on the different questionnaires assessed. | 6 weeks : before the first session of rTMS (vocal samples) and before and after the treatment (questionnaires)
  Coefficients of determination R² and average absolute errors between the scores predicted by the model and the actual scores obtained on the different PHQ-9, GAD-7, IADL, AIS and MAP-SR questionnaires.
Area under the curve of the different prediction models obtained, starting from pre-trained models on healthy subject databases. | 6 weeks : Before and after rTMS treatment
  Area under the curve of the different prediction models obtained, starting from pre-trained models on healthy subject databases.
Risk and coverage of the different prediction models obtained. | 6 weeks : After rTMS treatment
  Risk and coverage of the different prediction models obtained.
Comparison of the prediction models obtained with or without the use of advanced data encryption algorithms. | 6 weeks : After rTMS treatment
  Comparison of the areas under the curve of the different prediction models obtained with or without the use of advanced data encryption algorithms.

OTHER OUTCOMES:
Self-evaluation of depressive symptoms | 6 weeks : weekly
  PHQ-9 questionnaire
Generalised Anxiety Disorder | 6 weeks : weekly
  GAD-7 questionnaire
Athens Insomnia Scale | 6 weeks : before and after rTMS treatment
  AIS questionnaire
Instrumental Activities of Daily Living (autonomy) | 6 weeks : before and after rTMS treatment
  IADL
Motivation and Pleasure Scale - Self Report (anhedonia) | 6 weeks : before and after rTMS treatment
  MAP-SR
Social Network Index | before rTMS treatment
  SNI
Loneliness Scale | before rTMS treatment
  UCLA 3-Items
Simple physical activity questionnaire | 6 weeks : before and after rTMS treatment
  SIMPAQ

CONTACTS AND LOCATIONS:
Overall Officials: Fariba KABIRIAN, MD, Principal Investigator — France Chief Medical Officer, Clariane
Locations (9):
- France (9):
  - Clinique Inicea du Pays de Seine, Bois-le-Roi
  - Clinique Inicea La Mare O Dans, Les Damps
  - Clinique Inicea Villa des Roses, Lyon
  - Etablissement public de santé de Ville-Evrard, Neuilly-sur-Marne
  - Centre médical de psychiatrie NeuroStim Luxembourg, Paris
  - Centre médical de psychiatrie NeuroStim Etoile, Paris
  - Clinique Inicea Jeanne d'Arc Hopital Privé Parisien, Saint-Mandé
  - Centre montois de psychiatrie ambulatoire Inicea, Saint-Pierre-du-Mont
  - Centre Tourangeau de psychiatrie ambulatoire Inicea, Tours

IPD SHARING:
Plan to Share IPD: Undecided